CLINICAL TRIAL: NCT02065440
Title: The Effect of Ebastine/Pseudoephedrine on Subacute Cough :a Randomized Placebo-controlled Trial
Brief Title: The Effect of Ebastine/Pseudoephedrine on Subacute Cough
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-2011-65
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Cough
Keywords: Ebastine/Pseudoephedrine; subacute cough; upper airway cough syndrome
MeSH Terms: conditions — Cough; upper airway cough syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ebastine/Pseudoephedrine (Active Comparator): administration of ebastine/pseudoephedrine 1cap/day for 1 week.
  Interventions: Drug: Rhinoebastel
- placebo (Placebo Comparator): administration of placebo pill 1 cap/day for 1week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rhinoebastel — Rhinoebastel(ebastine 10mg/pseudoephedrine 120mg) 1 cap/day for 1 week unless progression or unacceptable toxicity develops.
  Arms: Ebastine/Pseudoephedrine
Drug: Placebo — Placebo 1 cap/day for 1 week unless progression or unacceptable toxicity develops
  Arms: placebo

SUMMARY:
To determine whether ebastine/pseudoephedrine is effective on subacute cough.

DETAILED DESCRIPTION:
1. Visit 0 week

   * Patients with subacute cough,area randomized to either ebastine/pseudoephedrine or placebo for 1 week.
   * The cough severity and quality of life were measure with VAS score and cough-specific quality-of-life questionnaire(CQLQ)
2. Visit 1 week check VAS score and CQLQ
3. Visit 4 weeks check VAS score and CQLQ

ELIGIBILITY:
Inclusion Criteria:

* patients with subacute cough(3-8 weeks)
* age: 20-70 years

Exclusion Criteria:

* Chest X-ray abnormality(+) as a probable cause of cough
* other explainable confirmed diagnosis(+) such as acute infectious disease
* Severe cough or cough complication which needs other anti-tussive agents.
* on ACEI
* with more than three hypertensive agents
* change of hypertension medication 3 months ago
* immunocompromized host
* relative or absolute contraindication for ebastine/pseudoephedrine

  1. hypersensitivity to ebastine/pseudoephedrine
  2. glaucoma
  3. moderate to severe hypertensive disease
  4. coronary heart disease
  5. hyperthyroidism
  6. moderate to severe liver disease
  7. benign prostate hyperplasia
  8. psychological problem
  9. Parkinson's disease
  10. on linezolid or supposed to use it.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Change of VAS score | 1 week later after administration of ebastine/pseudoephedrine or placebo

SECONDARY OUTCOMES:
Change of VAS score | 4 weeks later after administration of ebastine/pseudoephedrine or placebo
The proportion of patients with more than 50 percent decrease in VAS score | 1 week
Change of CQLQ score | 1week later after administration of ebastine/pseudoephedrine or placebo
Change of CQLQ score | 4 weeks later after administration of ebastine/pseudoephedrine or placebo
The adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Lee, MD, Study Chair — Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Seoul Metropolitan Government, Seoul National University Boramae Medical Center
Locations (1):
- Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Seoul Metropolitan Government, Seoul National University Boramae Medical Center, Seoul, Dongjak-Gu, South Korea